CLINICAL TRIAL: NCT01763151
Title: Comparison of Toric IOL Implantation and Opposite Clear Corneal Incision During Cataract Surgery to Correct Corneal Astigmatism
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Vienna Institute for Research in Ocular Surgery (Other)
Responsible Party: Principal Investigator, Prim. Prof. Dr. Oliver Findl, MBA, MD, MBA, Vienna Institute for Research in Ocular Surgery
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Viros_Askin
Record Dates: First submitted 2013-01-06; First posted 2013-01-08 (Estimated); Last update posted 2013-01-10 (Estimated); Status verified 2013-01

CONDITIONS: Cataract; Corneal Astigmatism
Keywords: cataract surgery, astigmatism, opposite clear corneal incision, toric IOL, IOL rotational stability
MeSH Terms: conditions — Cataract; Astigmatism

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- toric IOL (Active Comparator): aspherical, toric acrylic IOL (Lentis L-312T, Oculentis, Germany)
  Interventions: Device: toric IOL
- IOL combined with opposite clear corneal incision (OCCI) (Active Comparator): aspherical, acrylic IOL with OCCI
  Interventions: Procedure: IOL combined with opposite clear corneal incision (OCCI)

INTERVENTIONS:
Device: toric IOL — implantation of an aspheric, toric, acrylic IOL during cataract surgery
  Arms: toric IOL
Procedure: IOL combined with opposite clear corneal incision (OCCI) — aspherical, acrylic IOL with opposite clear corneal incision during cataract surgery
  Arms: IOL combined with opposite clear corneal incision (OCCI)

SUMMARY:
With increasing demands of patients concerning refractive outcome after cataract surgery, toric intraocular lenses (IOLs) that correct corneal astigmatism have been introduced more widely to cataract surgery. Originally toric IOLs were used mainly for patients with high degrees of astigmatism, especially after corneal surgical procedures such as penetrating keratoplasty. Since a couple of years, toric IOLs are available from numerous manufacturers to correct lower amounts of astigmatism which are much more prevalent with about 30% having a corneal astigmatism of 0.75D or more in the cataract population. This should result in less spectacle dependence of patients due to the astigmatic correction.

The alternative method to reduce corneal astigmatism as part of cataract surgery is to make incisions on the steeper axis of the cornea such as limbal relaxing incisions or an additional clear corneal incision opposite (OCCI) to the main cataract opening. These techniques are in use since more than 2 decades and are widely used in clinical routine. As with toric IOLs, precise alignment of the cuts with the axis of astigmatism is essential. The disadvantage of the incisional techniques is the variability of the effect between patients since it depends on factors such as the extent of scaring of the cuts after surgery as well as corneal thickness. The main advantage is the simplicity of the technique and the lower cost.

Aim of this study is to compare toric IOL implantation and opposite clear corneal incision during cataract surgery to correct corneal astigmatism.

ELIGIBILITY:
Inclusion Criteria:

* Cataract
* Age 21 and older
* Regular corneal astigmatism 1.0 up to 2.5 D
* written informed consent prior to surgery

Exclusion Criteria:

* Relevant other ophthalmic diseases such as: pseudoexfoliation, glaucoma, traumatic cataract corneal scars, and other co-morbidity that could affect capsule bag stability ( e.g. Marfan syndrome)
* Irregular corneal astigmatism on corneal topography

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2010-09; Primary Completion 2012-08 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Postoperative residual astigmatism | 9 months post-operatively

SECONDARY OUTCOMES:
uncorrected distance visual acuity (UDVA) | 9 months post-operatively

OTHER OUTCOMES:
postoperative IOL rotation | 3 months and 9 months post-operatively

CONTACTS AND LOCATIONS:
Locations (1):
- Vienna Institute for Research in Ocular Surgery (VIROS), Hanusch Hospital, Vienna, Austria